CLINICAL TRIAL: NCT01127282
Title: The Impact of Vitamin on the Clinical Course in Cases Infected by Novel H1N1 Influenza Virus A: a Randomized-controlled Trial
Brief Title: The Impact of Vitamin on the Clinical Course in Cases Infected by Novel H1N1 Influenza Virus A
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Chang-Hoon Lee, Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vitamin_H1N1
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: H1N1 Influenza
Keywords: influenza; vitamin; improvement of symptom
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — Vitamins; Vitamin A; Digestion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin (Experimental): Vitamin(vitamin A 15mg,C 500mg,E 400IU) 1T po for 5 days in addition to anti-viral agent and antipyretics
  Interventions: Drug: Vitamin (vitamin A 15 mg,C 500 mg, E 400IU)
- Control (Placebo Comparator): Placebo(digestive tablet) 1T po for 5 days in addition to anti-viral agent and antipyretics
  Interventions: Drug: Placebo (digestive tablet)

INTERVENTIONS:
Drug: Vitamin (vitamin A 15 mg,C 500 mg, E 400IU) — Vitamin (vitamin A 15 mg,C 500 mg, E 400IU) 1T po for 5 days in addition to anti-viral agent and antipyretics
  Arms: Vitamin
Drug: Placebo (digestive tablet) — Placebo (digestive tablet) 1T po for 5 days in addition to anti-viral agent and antipyretics
  Arms: Control

SUMMARY:
Influenza continues to inflict an important burden on health-care systems. The 2009 H1N1 influenza virus first appeared in Mexico and the United States in March and April 2009 and has swept the globe with unprecedented speed.

The aim of this study is to evaluate effect of supplement vitamin on the clinical course of patients with acute respiratory illness suspected novel H1N1 infection.

DETAILED DESCRIPTION:
Patients with acute respiratory illness randomized to control or vitamin groups. The patients completed questionnaire about their initial symptom scores. After 5 days of vitamin trial, patients were asked about their symptom by telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* Acute respiratory illness suspected H1N1 infection
* Acute febrile respiratory illness(BT > 37.8) and throat pain or cough or nasal congestion

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to vitamin A
* History of liver disease or renal disease
* Urinary stone disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
change of symptom score | 1 week after initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Lee, MD, Study Chair — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Locations (1):
- Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul Metropolitan Government, Seoul National University Boramae Medical Center, Seoul, South Korea